CLINICAL TRIAL: NCT00852709
Title: Phase I Dose-Escalation Trial of Clofarabine Followed by Escalating Doses of Fractionated Cyclophosphamide in Children With Relapsed or Refractory Acute Leukemias
Acronym: POE07-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0715; POE07-01
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Myelodysplastic Syndrome; Acute Myeloid Leukemia; Myeloproliferative Disorders; Acute Lymphocytic Leukemia; Acute Promyelocytic Leukemia; Acute Leukemia; Chronic Myelogenous Leukemia; Myelofibrosis; Chronic Myelomonocytic Leukemia; Juvenile Myelomonocytic Leukemia
Keywords: Myelodysplastic syndrome that has transformed to AML (AML/MDS); Treatment-related AML; AML evolving from myeloproliferative disorders (MPD); Acute lymphocytic leukemia (ALL); Acute promyelocytic leukemia (APL) refractory to arsenic therapy or retinoic acid therapy; Relapsed and/or refractory acute leukemia with progressive disease since last therapy; Chronic myelogenous leukemia (CML) in accelerated phase or blast crisis refractory to imatinib; High-risk MPD including myelofibrosis, chronic myelomonocytic leukemia (CMML, and relapsed or refractory juvenile myelomonocytic leukemia (JMML).
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Promyelocytic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myelomonocytic, Juvenile; Recurrence | interventions — Clofarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clofarabine — On Days 1, 2, and 3 and Days 8, 9, and 10 clofarabine will be administered by IVI 2 hours before each dose of cyclophosphamide
Drug: Cyclophosphamide — Single-agent cyclophosphamide will be administered by 2-hour IVI on Day 0 of cycle 1. On Days 1, 2, and 3 and Days 8, 9, and 10 clofarabine will be administered by IVI 2 hours before each dose of cyclophosphamide

SUMMARY:
This is a Phase I study designed to determine the MTD and assess the toxicity associated with clofarabine followed by fractionated cyclophosphamide in patients > 1 year of age or < 21 years of age with relapsed or refractory acute leukemias. There will be 25 to 35 patients enrolled. Cohorts of 3 to 6 patients each will receive escalated doses of clofarabine followed by fractionated cyclophosphamide until the MTD is reached. There will be no intra-patient dose escalation. Single-agent cyclophosphamide will be administered by 2-hour IVI on Day 0 of cycle 1. On Days 1, 2, and 3 and Days 8, 9, and 10 clofarabine will be administered by IVI 2 hours before each dose of cyclophosphamide (see the treatment schema below). A cycle is defined as 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 for adolescent/young adult patients.
* Lansky Performance Index > 50 for pediatric patients less than age 10 years.
* Laboratory values obtained < 7 days prior to receiving study treatment:
* Total bilirubin < 1.5 mg/dL unless elevated due to hemolysis. The conjugated serum bilirubin prior to study entry must be within the normal range.
* Aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 × upper limit of normal (ULN)
* Serum creatinine < 1.0 mg/dL in adolescent/young adults (patients 12 to 17 years of age). For pediatric patients with serum creatinine above the ULN, creatinine clearance > 90 ml/min/1.73m2 calculated using the Schwartz formula may be enrolled. Collected creatinine clearance may be substituted.

Patients 18 years and older (Adult population): Serum creatinine <1.0 mg/dL; if serum creatinine >1.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be >60 mL/min/1.73 m2

* Cardiac function must be normal per the institution normal as measured by echocardiogram (ECHO) within 7 days.
* Patients should have no evidence of myositis as detected by abnormal serum creatine kinase and/or myoglobin.

Exclusion Criteria:

* No chemotherapy, radiation, or major surgery within 2 weeks prior to first dose of study drug except for 5-azacytidine, thalidomide, hydroxyurea, imatinib (Gleevec), and interferon which must be discontinued at least 3 days before study entry and the patient should have recovered from the toxic side effects of such therapy. In the instance of progressive disease, anti-leukemia therapy may have been administered within the 2-week period as long but the subject should have recovered from the toxic effects of that therapy. Also, intrathecal therapy may be administered within the 2-week period for subjects with CNS disease.
* Patients who have had an allogeneic or autologous hematopoietic stem cell transplant.
* Patients must have discontinued all growth factors, except Procrit (epoetin), at least 1 week before study.
* Patients with known HIV positive status or AIDS.
* Patients with known active Hepatitis B, Hepatitis C or cirrhosis.
* History of severe coronary artery disease, including myocardial infarction within the previous 3 months, arrhythmias other than atrial flutter or fibrillation requiring medication, or uncontrolled congestive heart failure.
* Patients with active uncontrolled infection, fever of infection, or evidence for progressive disease by CT scans of the lungs, sinuses, or abdomen. Patients who are on antimicrobial therapy and stable, CT scans must have been stable for 4 weeks, may be enrolled but there must be no evidence of an active infection. Patients with fever due to leukemia may be enrolled.
* Pregnant or lactating patients. Female patients of childbearing potential must have a negative serum pregnancy test within 14 days before study entry.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-09-01 (Actual); Primary Completion 2009-11-20 (Actual); Study Completion 2009-11-20 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility, tolerability, toxicities, and MTD of clofarabine followed by fractionated cyclophosphamide in pediatric patients with relapsed or refractory acute leukemias. | 1 cycle

SECONDARY OUTCOMES:
To obtain preliminary descriptive data of the biologic and pharmacodynamic effects of clofarabine followed by fractionated cyclophosphamide on marrow and circulating leukemic blasts in pediatric patients with relapsed or refractory acute leukemias. | 1 cycle

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Colorado Health Sciences Center and The Children's Hospital, Aurora, Colorado
  - Pediatrix Hematology/Oncology University of Florida College of Medicine, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - M.D. Anderson Comprehensive Cancer Center, Houston, Texas
- Southern Alberta Children's Cancer Program, Calgary, Alberta, Canada